CLINICAL TRIAL: NCT00571233
Title: Identification of Biomarkers for Heart Failure in Children With Single Ventricle Physiology
Brief Title: Biomarker Study for Heart Failure in Children With Single Ventricle Physiology
Acronym: BHFSVP
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 2529
Record Dates: First submitted 2007-12-05; First posted 2007-12-11 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Tricuspid Atresia; Hypoplastic Left Heart Syndrome; Unbalanced AV Canal
Keywords: Single Ventricle; Congenital Heart Disease; Children; Fontan; Tricuspid Atresia; Hypoplastic Left Heart Syndrome; Heart Failure; Biomarkers; Single ventricle physiology such as:; unbalanced AV canal; Interested in patients both before and after Fontan Surgery
MeSH Terms: conditions — Tricuspid Atresia; Hypoplastic Left Heart Syndrome; Univentricular Heart; Heart Defects, Congenital; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Group one consists of children 1 month - 6 years old who have structurally normal hearts, no heart failure, and a patent ductus arteriosus (PDA).
- 2: Group two consists of children 1 month - 6 years old who have single ventricle physiology. Children with and without heart failure may participate.

SUMMARY:
The purpose of this study is to determine if children with heart disease where there is only one pumping chamber("ventricle") have proteins (biomarkers") in the blood that can be used to monitor the function of their heart.

DETAILED DESCRIPTION:
We will investigate whether levels of blood proteins in children with well-functioning hearts with one ("single") ventricle are similar to levels of these blood proteins in children with two ventricles. For children with hearts with a single ventricle, we will examine blood proteins at various levels of heart function. To assess blood protein levels, we will collect small (6 mL) samples of blood. Heart function will be determined by existing clinical scoring systems. Enrolled patients will receive an echocardiogram, which is a dynamic ultrasound picture of the beating heart.

ELIGIBILITY:
Inclusion Criteria:

* Children with a structurally normal heart and a patent ductus arteriosus.
* Children with single ventricle physiology.

Exclusion Criteria:

* Children must not have chromosomal abnormalities. Small deletions, such as that which produces DiGeorge syndrome, are permissible.
* Children with acute intercurrent non-cardiac inflammatory illness (such as post-operative wound infection) are ineligible, as such conditions may cause elevated blood levels of the proteins under study.

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients presenting to the UCSF Pediatric Heart Center.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2007-02; Primary Completion 2011-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Heart failure, as assessed by clinical scoring systems. | Cross-sectional. We will obtain blood samples and assess for heart failure (function) concurrently when patients present to the Pediatric Heart Center

SECONDARY OUTCOMES:
Echocardiographic indices. | Cross-sectional

CONTACTS AND LOCATIONS:
Overall Officials: Harold Bernstein, MD, PhD, Principal Investigator — UCSF Pediatric Cardiology
Locations (1):
- Pediatric Heart Center, University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Result] Shah A, Feraco AM, Harmon C, Tacy T, Fineman JR, Bernstein HS. Usefulness of various plasma biomarkers for diagnosis of heart failure in children with single ventricle physiology. Am J Cardiol. 2009 Nov 1;104(9):1280-4. doi: 10.1016/j.amjcard.2009.06.046. PMID 19840577
- [Result] Lowenthal A, Shah A, Bernstein HS. Letter by Lowenthal et al regarding article, "BNP levels predict outcome in pediatric heart failure patients: post hoc analysis of the Pediatric Carvedilol Trial". Circ Heart Fail. 2010 Nov;3(6):e32; author reply e33. doi: 10.1161/CIRCHEARTFAILURE.110.958470. No abstract available. PMID 21081737
- [Result] Lowenthal A, Camacho BV, Lowenthal S, Natal-Hernandez L, Liszewski W, Hills NK, Fineman JR, Bernstein HS. Usefulness of B-type natriuretic peptide and N-terminal pro-B-type natriuretic peptide as biomarkers for heart failure in young children with single ventricle congenital heart disease. Am J Cardiol. 2012 Mar 15;109(6):866-72. doi: 10.1016/j.amjcard.2011.10.049. Epub 2011 Dec 22. PMID 22196786
- See also: Usefulness of Various Plasma Biomarkers for Diagnosis of Heart Failure in Children with Single Ventricle Physiology — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2791782/?tool=pubmed
- See also: Letter by Lowenthal et al regarding article, "BNP levels predict outcome in pediatric heart failure patients: post hoc analysis of the Pediatric Carvedilol Trial" — http://www.ncbi.nlm.nih.gov/pubmed/21081737
- See also: Usefulness of B-Type Natriuretic Peptide and N-Terminal Pro-B-Type Natriuretic Peptide as Biomarkers for Heart Failure in Young Children With Single Ventricle Congenital Heart Disease — http://www.ncbi.nlm.nih.gov/pubmed/22196786